CLINICAL TRIAL: NCT02555579
Title: Use of Dietary Protein and Free Fruits and Vegetables to Improve Metabolic Control Among Teens and Adults With Phenylketonuria: A Mixed Methods Approach
Brief Title: Simplified Diet Approach in Phenylketonuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0451-15-EP
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary Protein Counting & Free Fruits & Vegetables (Experimental): Subjects will be educated on new simplified diet approach and phenylalanine levels will be monitored for 1 year, and will be compared to 12 months prior to study enrollment
  Interventions: Behavioral: Dietary Protein Counting and Free Fruits and Vegetables

INTERVENTIONS:
Behavioral: Dietary Protein Counting and Free Fruits and Vegetables — Subjects will be educated on new simplified diet approach and phenylalanine levels will be monitored for 1 year, and will be compared to 12 months prior to study enrollment

SUMMARY:
This is a study to determine if a simplified protein counting system, including the free usage of fruits and vegetables low in phenylalanine, will improve the metabolic control in teens and adults with phenylketonuria (PKU).

Anybody with a positive diagnosis of PKU, between the ages of 13-65 years will be invited to participate in this study.

Subjects will be educated on the simplified system upon enrollment, and historical phenylalanine (Phe) levels will be used for comparison. Subjects will also be asked about their attitudes towards their current Phe counting system.

DETAILED DESCRIPTION:
This is a study to determine if a simplified protein counting system, including the free usage of fruits and vegetables low in phenylalanine, will improve the metabolic control in teens and adults with phenylketonuria (PKU).

Anybody with a positive diagnosis of PKU, between the ages of 13-65 years will be invited to participate in this study.

Subjects will be educated on the simplified system upon enrollment, and historical phenylalanine (Phe) levels will be used for comparison. Subjects will also be asked about their attitudes towards their current Phe counting system.

Upon enrollment, a 3-day food record and Phe levels over the past 12 months will be collected. Demographic information will be asked, as well as questions regarding their current Phe counting system. Patients will be educated on the new counting system, stressing 3 key principles: 1) free use of fruits and vegetables, low in protein, 2) protein counting as a simpler version of Phe counting, including reinforcement of label reading, and 3) daily use of PKU formula for enhanced nutrient and protein intake. Patients will be given written educational tools to reinforce this new method.

At the end of the 12 months, subjects will be asked to provide a 3-day food record, and questions will be asked about their attitudes toward the use of the new simplified system.

Phenylalanine levels from the 12-month study period will be used to compare with historical data.

ELIGIBILITY:
Inclusion Criteria:

1. Positive diagnosis of PKU
2. Males and females >13 year of age
3. Currently on phenylalanine-restricted diet

Exclusion Criteria:

1. Any woman planning, or becoming pregnant during study duration
2. Any patient who starts Kuvan during the study, as Kuvan lowers phenylalanine levels in some patients.
3. Any patient currently enrolled in other research studies (Prism 301/302 Protocol; Institutional Review Board Protocol # 376-13-FB)

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Metabolic Control in Teens and Adults with PKU | 12 months
  phenylalanine levels

SECONDARY OUTCOMES:
attitudes towards simplified diet approach | 12 months
  qualitative data collection

CONTACTS AND LOCATIONS:
Overall Officials: Jill C Skrabal, PhD, Principal Investigator — University of Nebraska
Locations (4):
- United States (4):
  - Monroe-Meyer Insititute, Omaha, Nebraska
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - Nebraska Medicine, Midtown Health Center, Omaha, Nebraska
  - Unversity of Nebraska Medical Center, Omaha, Nebraska